CLINICAL TRIAL: NCT01237457
Title: 177Lutetium-DOTA-Octreotate Therapy in Somatostatin Receptor-Expressing Neuroendocrine Neoplasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ebrahim S Delpassand (Other)
Collaborators: Excel Diagnostics and Nuclear Oncology Center (Other)
Responsible Party: Sponsor-Investigator, Ebrahim S Delpassand, Chairman and Medical Director, Excel Diagnostics and Nuclear Oncology Center
Organization: Excel Diagnostics and Nuclear Oncology Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 78,256
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients with somatostatin receptor-expressing neuroendocrine neoplasms will receive up to 200 mCi of 177Lu-DOTATATE every 6-11 weeks, preferably 6-9 weeks to a cumulative dose of 800 mCi.
  Interventions: Drug: 177Lu-DOTATATE

INTERVENTIONS:
Drug: 177Lu-DOTATATE — Patients will receive 200mCi dose of 177Lu Dotatate

SUMMARY:
This is a phase II treatment protocol evaluating 177Lu-DOTATATE therapy for somatostatin receptor-expressing cancers including, but not limited to, those arising from the neural crest and involving such organs as the lungs, breast, gastrointestinal tract, skin, and endocrine (examples: pheochromocytoma, medullary carcinoma of the thyroid, non-radioiodine avid differentiated thyroid cancer, melanoma, renal cell, Merkel cell, paraganglioma, small cell lung, Carcinoid, and pancreatic islet cell malignancies).

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven Gastroenteropancreatic (GEP tumors including bronchial carcinoids)
* Presence of somatostatin-receptors on the known tumor lesions demonstrated by OctreoScan within 6 months of the first dose of radiolabelled octreotate therapy. The uptake on the OctreoScan should be at least as high as normal liver uptake on planar imaging.
* Life Expectancy greater than 12 weeks.
* Serum creatinine ≤ 150 µmol/liter or 1.7 mg/dL and a measured creatinine clearance (or measured GFR using plasma clearance methods, not gamma camera based) of ≥ 50ML/min.
* Hemoglobin (Hgb) concentration ≥ 5.5 mmol/L (≥ 8.9 g/dL); WBC ≥ 2*109/L (2000/mm3); platelets ≥ 100*109/L (100*103/mm3).
* Total Bilirubin ≤ 3X UNL.
* Serum Albumin > 30g/L or serum albumin ≤ 30g/L but normal prothrombin time.
* All patients must have a Karnofsky performance status of at least 60%
* Patients must be greater than 18 years of age. Patients younger than 18 years will be presented to FDA for compassionate use on a case by case basis

Exclusion Criteria:

* Possible surgery with curative intent.
* Surgery, radiotherapy, chemotherapy or other investigational therapy within 3 months of the start of therapy.
* Patients with known brain metastases unless these metastases have been treated and stabilized for at least 6 months prior to study start. Patients with a history of brain metastases must have a head CT with contrast to document stable disease prior to study start.
* Uncontrolled congestive heart failure.
* Any subject who is taking concomitant medications which decrease renal function (such as aminoglycoside antibiotics).
* Any subject receiving therapy with somatostatin analogues, unless the dose has been stable for at least 3 months prior to the first cycle in this study and the disease status during these 4 months has been documented by modified RECISTS criteria as described in this study
* Any subject receiving therapy with short acting somatostatin analogues in whom these analogues cannot be interrupted for 12 hours before and 12 hours after the administration of the radio labelled somatostatin analogues, or any subject who receives therapy with long-acting somatostatin analogues in whom these analogues cannot be interrupted for at least 6 weeks before the administration of the radio labeled somatostatin analogues, unless the uptake on the Octreoscan during continued somatostatin analogue medication is at least as high as normal liver uptake on planar imaging.
* In patients with unusual hematological parameters, including an increased MCV (>105fL), and especially in those who had previous chemotherapy, the advice of a hematologist should be sought for adequate further work-up.
* Subjects with another significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with completion of the study.
* Prior radiation therapy to more than 25% of the bone marrow.
* Female patients who are pregnant, lactating or women of childbearing potential not willing to practice effective contraceptive techniques during the study period and for 60 days (10 half lives of 177Lu after the last treatment, or male patients who have female partners of childbearing potential not willing to practice abstinence or effective contraception, during the study period and for 60 days after the last treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2010-10-27 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Progression Free survival | one year after completion of last treatment cycle
  Overall response will be determined by Progression Free Survival (PFS). PFS will be calculated as a function of time from start of therapy to time of overall disease progression. Patients will be censored at the date of last contact

SECONDARY OUTCOMES:
Dose limiting toxicity | one year after completion of the fourth cycle of treatment
  Patients will be monitored for dose toxicity according to NCI guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim S Delpassand, M.D, Principal Investigator — Excel Diagnostics and Nuclear Oncology Center
Locations (1):
- Excel Diagnostics and Nuclear Oncology Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No